CLINICAL TRIAL: NCT02004314
Title: Chloroquine as a Modulator of T Cell Immune Activation to Improve CD4 Recovery in HIV-infected Participants Receiving Antiretroviral Therapy: A Proof-of-concept Study
Brief Title: Chloroquine as a Modulator of T Cell Immune Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTN 246
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: HIV
Keywords: Chloroquine; T cell immune activation; CD4 recovery; HIV
MeSH Terms: interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chloroquine (Other): This will be a single arm, pilot study with each subject as his/her own control. The study will last 44 weeks, with 8 weeks observation period on ART alone to assess stability of activated CD8CD38 T cells, followed by 24 weeks chloroquine treatment with ART and a 12-week follow-up period on ART alone. Twenty ART treated patients will be recruited. To maximize chances of demonstrating a treatment effect, the chloroquine will be administrated for 24 weeks.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine

SUMMARY:
This study will evaluate the effect of chloroquine in individuals infected with HIV. Researchers will aim to determine if chloroquine treatment in participants whose viral loads are suppressed on combination antiretroviral therapy (ART), results in improved immune activation and CD4 cell recovery.

The study will recruit 20 individuals and will last approximately 44 weeks. Eligible participants will receive an oral dose of chloroquine (250 mg) once daily from week 8 through week 32. All participants will be asked to have rectal biopsy samples (week 0 and week 32) to study T cell immune activation in the mucosa rectal site.

DETAILED DESCRIPTION:
Clinical data has identified chloroquine as a potential modulator of immune activation. The study's dose of chloroquine is the same as the dose recommended for patients having autoimmune diseases. In these autoimmune cases, a daily dose of chloroquine at 250 mg for 12 weeks has shown improvement in symptoms and decreases in inflammatory cytokines synthesis and a reduction in TLR -mediated immune activation. Study findings could help provide information about where and under what circumstances chloroquine treatment may reduce T cell activation and help restore circulating CD4 T cells.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection by Western Blot, EIA assays or viral load assay.
* Aged between 18 and 65 years.
* Viral load less than 50 copies per ml for at least the previous 36 weeks.
* CD4 cell count less than or equal to 350 cells per litre.
* On stable ART
* Vital signs, physical examination and laboratory results do not exhibit evidence diseases such as advanced cirrhosis or advanced liver
* Karnofsky performance status greater than or equal to 80 per cent.
* Participant does not require and agrees not to take, for the duration of the study, any medication that is contraindicated with chloroquine.
* Able to give informed consent.

Exclusion Criteria:

* Active AIDS events in the last 3 months
* Co-infection with active hepatitis B or C virus.
* Current use or use within four weeks prior to the baseline visit, of cytotoxic agents, systemic corticosteroids or any immuno-modulatory agents.
* Current use within four weeks prior to the chloroquine therapy the following medications: methadone, chlorpromazine, cimetidine, cyclosporin, methotrexate and penicillanime.
* Psychiatric or cognitive disturbance or illness that could preclude compliance with the study.
* Patient with clinically significant hemophilia and Von-Willebrand disease and any severe bleeding disorder.
* Experimental HIV immune based therapy within 6 months of screening visit.
* Allergic reaction to chloroquine.
* A history of retinitis or any retinal problem.
* Subjects with G6PD deficiency, porphyria, psoriasis, cirrhosis, hearing deficiency (including tinnitus), myopathy and cardiomyopathy.
* Pregnant and breast-feeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The expression of CD38 on CD8 circulating T cells | 44 weeks, with 8 weeks observation period on ART alone to assess stability of activated CD8CD38 T cells, followed by 24 weeks chloroquine treatment with ART and a 12-week follow-up period on ART alone
  To assess whether the expression of CD38 on CD8 circulating T cells will be reduced and whether circulating CD4 T cell recovery will be enhanced after 24 weeks of chloroquine treatment in adults whose HIV replication is suppressed by ART.

SECONDARY OUTCOMES:
Safety of chloroquine treatment measured by adverse events, hematology and serum chemistries and Amsler grid test. | 44 weeks, with 8 weeks observation period on ART alone to assess stability of activated CD8CD38 T cells, followed by 24 weeks chloroquine treatment with ART and a 12-week follow-up period on ART alone
  Safety of chloroquine treatment measured by adverse events, hematology and serum chemistries and Amsler grid test

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Chest Institute, McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Routy JP, Angel JB, Patel M, Kanagaratham C, Radzioch D, Kema I, Gilmore N, Ancuta P, Singer J, Jenabian MA. Assessment of chloroquine as a modulator of immune activation to improve CD4 recovery in immune nonresponding HIV-infected patients receiving antiretroviral therapy. HIV Med. 2015 Jan;16(1):48-56. doi: 10.1111/hiv.12171. Epub 2014 Jun 2. PMID 24889179